CLINICAL TRIAL: NCT02099630
Title: Functional and Metabolic Changes in the Course of Antidepressive Treatment
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Simone Grimm, Research Fellow, Charite University, Berlin, Germany
Other Study IDs: EMOKET-103/13
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will investigate functional and metabolic changes in the course of antidepressive treatments.

The investigators will apply different imaging methods to investigate the effects of antidepressive interventions on resting state neural activity, functional activation during cognitive and emotional stimulation, neurotransmitter concentrations as well as concentrations of brain- derived neurotrophic factor.

DETAILED DESCRIPTION:
The study will investigate functional and metabolic changes in the course of antidepressive treatments.

The investigators will apply different imaging methods to investigate the effects of antidepressive interventions on resting state neural activity, functional activiation during cognitive and emotional stimulation, neurotransmitter concentrations as well as concentrations of brain- derived neurotrophic factor.

The investigators hypothesize that antidepressive interventions modulate the excitatory glutamatergic system and thereby increase either the concentration of glutamate or the glutamate/ glutamine ratio. These metabolic changes are accompanied by altered functional activation in medial and lateral prefrontal areas during emotional and cognitive stimulation, respectively. After longterm treatment, excitatory glutamate and inhibitory gamma-aminobutyric acid concentrations adapt to a new homeostatic level which is reflected in antidepressive response or remission of symptoms. The investigators assume that the levels of glutamate and gamma-aminobutyric acid determine the amplitude of BOLD responses during emotional and cognitive stimulation. Furthermore, the investigators hypothesize that the plasma concentration of brain- derived neurotrophic factor might be a predictor for therapy response and changes in the course of treatment.

With our protocol we adhere to the rules of good scientific practice and observe all relevant laws, regulations and guidelines that pertain to the project. The investigators' study is in compliance with the Declaration of Helsinki and approved by the local ethics committee. Storage of data is in accordance with german privacy laws.

ELIGIBILITY:
Inclusion Criteria:

* age 18- 65 years
* current depressive episode
* males and females
* Intelligence quotient > 80
* written informed consent

Exclusion Criteria:

* neurological or psychiatric disease other than major depressive disorder
* metal implants, pacemaker, intracranial clips
* agoraphobia
* history of serious head injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: depressive patients from a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2019-11 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in neurotransmitter concentrations (glutamate, glutamine, gamma-aminobutyric acid) from baseline to response to antidepressive intervention | Neurotransmitter concentrations will be measured at baseline (T0), after the first antidepressive intervention (T1; 24- 48 hrs. after baseline measurement) and after patients show response or remission of symptoms (T2; an expected average of 2- 4 weeks)
  Neurotransmitter concentrations will be measured at 3 timepoints (at baseline, after the first antidepressive intervention and after patients show response or remission of symptoms). Measurements will show whether antidepressive interventions modulate the excitatory glutamatergic system and thereby increase either the concentration of glutamate or the glutamate/ glutamine ratio. After longterm treatment, excitatory glutamate and inhibitory gamma-aminobutyric acid concentrations are hypothesized to adapt to a new homeostatic level which is reflected in antidepressive response or remission of symptoms.

SECONDARY OUTCOMES:
Change in neuronal activation patterns from baseline to response to antidepressive intervention | Measurements will be conducted at baseline (T0), after the first antidepressive intervention (T1; 24- 48 hrs. after baseline measurement) and after patients show response or remission of symptoms (T2; an expected average of 2- 4 weeks)
  Neuronal activation patterns will be measured at 3 timepoints (at baseline, after the first antidepressive intervention and after patients show response or remission of symptoms). Measurements will show whether antidepressive interventions modulate resting state neural activity and functional activiation during cognitive and emotional stimulation. We expect changes in neurotransmitter concentrations to be accompanied by altered functional activation in medial and lateral prefrontal areas during emotional and cognitive stimulation, respectively. Furthermore, levels of glutamate and gamma-aminobutyric acid are hypothesized to determine the amplitude of BOLD responses during emotional and cognitive stimulation.

OTHER OUTCOMES:
Change in brain- derived neurotrophic factor concentration from baseline to response to antidepressive intervention | Measurements will be conducted at baseline (T0), after the first antidepressive intervention (T1; 24- 48 hrs. after baseline measurement) and after patients show response or remission of symptoms (T2; an expected average of 2- 4 weeks)
  Brain- derived neurotrophic factor concentrations will be measured at 3 timepoints (at baseline, after the first antidepressive intervention and after patients show response or remission of symptoms). Measurements will show whether the plasma concentration of brain- derived neurotrophic factor might be a predictor for therapy response and changes in the course of treatment.

REFERENCES:
- [Derived] Herrera-Melendez A, Stippl A, Aust S, Scheidegger M, Seifritz E, Heuser-Collier I, Otte C, Bajbouj M, Grimm S, Gartner M. Gray matter volume of rostral anterior cingulate cortex predicts rapid antidepressant response to ketamine. Eur Neuropsychopharmacol. 2021 Feb;43:63-70. doi: 10.1016/j.euroneuro.2020.11.017. Epub 2020 Dec 11. PMID 33309459
- [Derived] Basso L, Bonke L, Aust S, Gartner M, Heuser-Collier I, Otte C, Wingenfeld K, Bajbouj M, Grimm S. Antidepressant and neurocognitive effects of serial ketamine administration versus ECT in depressed patients. J Psychiatr Res. 2020 Apr;123:1-8. doi: 10.1016/j.jpsychires.2020.01.002. Epub 2020 Jan 16. PMID 31981856
- [Derived] Gartner M, Aust S, Bajbouj M, Fan Y, Wingenfeld K, Otte C, Heuser-Collier I, Boker H, Hattenschwiler J, Seifritz E, Grimm S, Scheidegger M. Functional connectivity between prefrontal cortex and subgenual cingulate predicts antidepressant effects of ketamine. Eur Neuropsychopharmacol. 2019 Apr;29(4):501-508. doi: 10.1016/j.euroneuro.2019.02.008. Epub 2019 Feb 26. PMID 30819549